CLINICAL TRIAL: NCT01586702
Title: Intensified Secondary Prevention Intending a Reduction of Recurrent Events in TIA and Minor Stroke Patients (INSPiRE-TMS) A Randomized Trial Comparing a Patient Centered Support Program Versus Conventional Car
Brief Title: Intensified Secondary Prevention Intending a Reduction of Recurrent Events in TIA and Minor Stroke Patients
Acronym: INSPiRE-TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Technical University of Munich (Other); University of Erlangen-Nürnberg Medical School (Other); Praxis für Neurologie und Psychiatrie am Prinzregentenplatz, München (Unknown); Technische Universität Berlin (Other); Aarhus University Hospital (Other); Klinikum Ludwigshafen (Other); Vivantes Auguste-Viktoria-Klinikum (Unknown); Vivantes Clinic Neukölln (Other)
Responsible Party: Principal Investigator, Heinrich J Audebert, Head of Neurology at Campus Benjamin Franklin, Clinical Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EA2/084/11
Record Dates: First submitted 2012-04-23; First posted 2012-04-27 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Mini-Stroke
Keywords: Stroke, TIA, secondary prevention, support program, multifactorial intervention
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular care (No Intervention): Consisting of structured information given at hospital discharge regarding stroke etiology and recommended secondary prevention plus regular outpatient care by general practitioners or family doctors.
- Support program (Active Comparator): In addition to regular care: Up to 8 appointments in outpatient clinics. Results of risk factor measurements and assessed adherence to medical recommendations are shared with the patients. In case that a patients fails to meet target values, preventive measures will be modified directly or via recommendation to GPs / family doctors. Patients are also offered assistance in finding appropriate physical activities or smoking cessation programs.
  Interventions: Behavioral: Patient centered structured support program

INTERVENTIONS:
Behavioral: Patient centered structured support program — Behavioural: Structured support program
  Program with up to 8 outpatient appointments focusing on:
  * Measurement of risk factors
  * Assessment of medication intake
  * Monitoring of antithrombotic therapy
  * Joint agreement of an individual target plan
  Target values for risk factors:
  * Blood pressure < 140/85 mmHg (<130/80 in diabetics), normal circadian profile
  * HbA1c <7.5%
  * Nicotine abstinence
  * LDL < 100mg/dl (< 70mg/dl in high risk patients)
  * Physical activity ≥ 30min >2 x / week
  Targets for pharmaceutical treatment:
  * Platelet inhibitors for strokes / TIA of arterial etiology
  * Combined platelet inhibition over 3 months in symptomatic intra- or extracranial stenosis
  * Cumarins (INR 2-3) or new oral anticoagulants in AF patients
  * Statin treatment in patients with LDL >100mg/dl
  Intervention strategies:
  • According to Motivational Interviewing
  Other Names: Intensified secondary prevention
  Arms: Support program

SUMMARY:
Patients after TIA or Stroke are at high risk of experiencing a new stroke or myocardial infarction. Poor adherence to evidence based secondary prevention regimens is frequently seen. Support programs for patients may not only improve adherence to recommended therapies but also reduce the recurrence rate of stroke and heart attack. The investigators hypothesize that compared to regular care, a structured and patient centered secondary prevention program will lead to a relative risk reduction of at least 28% of recurrent vascular events.

DETAILED DESCRIPTION:
Although effective methods of secondary prevention after stroke or TIA are available, adherence to recommended evidence-based treatments is often poor. Programs for supported secondary prevention after cerebrovascular events with improved health education are promising but have not been evaluated regarding recurrent event reduction so far.

A prospective randomized trial has been started to assess the effectiveness of a patient centered structured support program intending a reduction of recurrent vascular events. Usual care consists of structured information given at discharge as well as regular outpatient care by general practitioners. The support program additionally employs a stepwise intensified support program with up to eight appointments over two years in outpatient clinics. Results of risk factor measurements and assessed adherence to medical recommendations are shared with the patients. They are also offered assistance in finding appropriate physical activities or smoking cessation programs.

Patients are randomized to regular care or regular care plus support program and will be followed-up until the total number of 317 primary endpoints has been reached. The composite primary endpoint consists of stroke, major coronary event and vascular death.

ELIGIBILITY:
Inclusion Criteria:

* Acute cerebrovascular event (either TIA or minor Stroke within 14 days before study inclusion) according to the following definitions:
* TIA (clinical restitution within 24 hours and ABCD2-Score ≥3) or visible DWI-lesion in MRI
* Minor stroke (mRankin ≤2 at time of inclusion)
* Patients with at least one of the following treatable risk factors:
* Arterial Hypertension
* Diabetes mellitus
* Atrial Fibrillation
* Smoking
* Written informed consent prior to study inclusion
* Realistic perspective in keeping the outpatient appointments

Exclusion Criteria:

* Distance from home to study center not in suitable range for keeping the outpatient appointments
* cognitive impairment jeopardizing adherence to the support program
* Modified Rankin Score >2 at time of study inclusion
* Malignant disease with life expectancy of less than 3 years
* relevant alcohol or other substance abuse (except for nicotine)
* Stroke or TIA etiology without options for evidence based secondary prevention (e.g. dissection or vasculitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2082 (Actual)
Dates: Start 2011-09; Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Major vascular event consisting of nonfatal stroke, nonfatal major coronary event and vascular death | Up to 6 years from inclusion
  Stroke: Acute (focal-) neurological syndrome, caused by brain infarction or intracerebral hemorrhage Major coronary event:Including instable Angina pectoris, STEMI and non-STEMI Vascular death: Caused by stroke (within 30 days of event), or major coronary event (within 7 days of event), or non-cerebral hemorrhage, or by peripheral arterial disease 30 days after vascular event or vascular intervention (intraarterial or surgical), or by pulmonary embolism or sudden death if death occurs within 24 hours in a patients with previously stable and healthy state if no non-vascular cause is documented

SECONDARY OUTCOMES:
Non vascular death | Participants will be followed-up for an average of approximately 3.5 years
Other vascular diseases leading to hospital admission (excl. primary outcome measure) | Participants will be followed-up for an average of approximately 3.5 years
  Consisting of TIA, Angina pectoris, PAD with vascular intervention
All hospital admissions with vascular intervention (intraarterial or surgical) | Participants will be followed-up for an average of approximately 3.5 years
Bleedings | Participants will be followed-up for an average of approximately 3.5 years
  All bleedings leading to therapeutic intervention (categorized according to GUSTO definitions)
Level of dependency | Up to 6 years from inclusion
  Assessment according to modified Rankin Score and level of care (German care insurance)
All hospital admissions | Participants will be followed-up for an average of approximately 3.5 years
Days alive and at home | Participants will be followed-up for an average of approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich J Audebert, MD, Principal Investigator — Center for Stroke Research, Charité Universitaetsmedizin Berlin
Locations (1):
- Dept. of Neurology, Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Stegemann A, Rios AS, Khalil A, Grittner U, Temuulen U, Ganeshan R, Braemswig TB, Horn A, Ihl T, Audebert HJ, Kufner A, Endres M. Neuroimaging Correlates of Post-Stroke Pain After Ischemic Stroke: Secondary Analysis of the INSPiRE-TMS Trial. medRxiv [Preprint]. 2025 Aug 11:2025.08.07.25333248. doi: 10.1101/2025.08.07.25333248. PMID 40832386
- [Derived] Ihl T, Ahmadi M, Laumeier I, Steinicke M, Ferse C, Klyscz P, Endres M, Hastrup S, Poppert H, Palm F, Kandil FI, Weber JE, von Weitzel-Mudersbach P, Wimmer MLJ, Audebert HJ. Patient-Centered Outcomes in a Randomized Trial Investigating a Multimodal Prevention Program After Transient Ischemic Attack or Minor Stroke: The INSPiRE-TMS Trial. Stroke. 2022 Sep;53(9):2730-2738. doi: 10.1161/STROKEAHA.120.037503. Epub 2022 Jun 15. PMID 35703097
- [Derived] Ahmadi M, Laumeier I, Ihl T, Steinicke M, Ferse C, Endres M, Grau A, Hastrup S, Poppert H, Palm F, Schoene M, Seifert CL, Kandil FI, Weber JE, von Weitzel-Mudersbach P, Wimmer MLJ, Algra A, Amarenco P, Greving JP, Busse O, Kohler F, Marx P, Audebert HJ. A support programme for secondary prevention in patients with transient ischaemic attack and minor stroke (INSPiRE-TMS): an open-label, randomised controlled trial. Lancet Neurol. 2020 Jan;19(1):49-60. doi: 10.1016/S1474-4422(19)30369-2. Epub 2019 Nov 7. PMID 31708447
- [Derived] Leistner S, Michelson G, Laumeier I, Ahmadi M, Smyth M, Nieweler G, Doehner W, Sobesky J, Fiebach JB, Marx P, Busse O, Kohler F, Poppert H, Wimmer ML, Knoll T, Von Weitzel-Mudersbach P, Audebert HJ. Intensified secondary prevention intending a reduction of recurrent events in TIA and minor stroke patients (INSPiRE-TMS): a protocol for a randomised controlled trial. BMC Neurol. 2013 Jan 24;13:11. doi: 10.1186/1471-2377-13-11. PMID 23347503
- [Derived] Leistner S, Benik S, Laumeier I, Ziegler A, Nieweler G, Nolte CH, Heuschmann PU, Audebert HJ. Secondary prevention after minor stroke and TIA - usual care and development of a support program. PLoS One. 2012;7(12):e49985. doi: 10.1371/journal.pone.0049985. Epub 2012 Dec 17. PMID 23284630